CLINICAL TRIAL: NCT04698824
Title: Hypnose en médecine Interne
Brief Title: Hypnosis in Internal Medecine
Acronym: HypnoMedIn
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Groupe Hospitalier Mutualiste de Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A03469-30
Record Dates: First submitted 2021-01-04; First posted 2021-01-07 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Hypnosis; Autoimmune Diseases; Medically Unexplained Symptoms
Keywords: internal medicine; survey; qualitative; impact of hypnosis
MeSH Terms: conditions — Autoimmune Diseases; Medically Unexplained Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Hypnosis session — At least one session of hypnosis in the internal medicine unit at the hospital "Groupe Hospitalier Mutualiste de Grenoble"

SUMMARY:
Description of the short and long-term impact of hypnosis sessions for patient having benefited from at least one hypnosis session in internal medicine at the french hospital "Groupe Hospitalier Mutualiste de Grenoble", with the help of a qualitative survey made by phone.

DETAILED DESCRIPTION:
The practice of hypnosis has experienced a recent boom in medicine, with a multiplication of its fields of action. Regarding internal medicine, the influence of the psyche on the immune system makes the use of hypnosis particularly relevant for autoimmune diseases. Medically unexplained symptoms (another important field of internal medicine) are also strongly psychosomatic and thus susceptible to hypnosis. The hypothesis is thus made that hypnosis can bring multiple benefits to internal medicine patients.

The main objective of this study is to describe the short and long-term impact of hypnosis sessions for patient having benefited from at least one hypnosis session in internal medicine at the french hospital "Groupe Hospitalier Mutualiste de Grenoble", with the help of a qualitative survey made by phone.

Moreover retrospective medical data concerning these patients will be collected to determine their medical history, their main symptoms et reasons to use hypnosis.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients who had at least one hypnosis session in internal medicine at the hospital "Groupe Hospitalier Mutualiste de Grenoble" between 08/28/2015 (date of the very first hypnosis consultation in internal medicine) and 03/17/2020 (date of confinement due to Covid19 in France)

Exclusion Criteria:

* Patient who had a hypnosis session, but who is not followed for a pathology in internal medicine or in internal medicine with a pneumological orientation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who had at least one hypnosis session in internal medicine at the hospital "Groupe Hospitalier Mutualiste de Grenoble" between 08/28/2015 (date of the very first hypnosis consultation in internal medicine) and 03/17/2020 (date of confinement due to Covid19 in France)
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Description of the short and long-term impact of hypnosis sessions thanks to a qualitative phone survey | Assessed only once. Phone call will be performed between march 2021 and June 2021
  Improvement in symptoms and quality of life, assessed thanks to a qualitative phone survey by 5-levels Likert scales

SECONDARY OUTCOMES:
Assessment of the reasons for patient satisfaction / dissatisfaction | Assessed only once. Phone call will be performed between march 2021 and June 2021
  Qualitative description by an open question in the phone survey
Description of the characteristics of these patients and of the hypnosis sessions | At inclusion
  Patients'characteristics described in medical records

CONTACTS AND LOCATIONS:
Overall Officials: Maxime LUGOSI, PhD, Principal Investigator — CHU Grenoble Alpes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lugosi M, Sacre K, Lidove O, Chauveheid MP, Brihaye B, Laissy JP, Chauchard M, Papo T. [Long-term follow-up of a French cohort of retroperitoneal fibrosis]. Rev Med Interne. 2013 Oct;34(10):591-9. doi: 10.1016/j.revmed.2013.02.002. Epub 2013 Mar 14. French. PMID 23498668
- [Background] Lugosi M, Alberti C, Zahar JR, Garrouste M, Lemiale V, Descorps-Desclere A, Ricard JD, Goldgran-Toledano D, Cohen Y, Schwebel C, Vesin A, Timsit JF, Azoulay E. Aspergillus in the lower respiratory tract of immunocompetent critically ill patients. J Infect. 2014 Sep;69(3):284-92. doi: 10.1016/j.jinf.2014.04.010. Epub 2014 Jun 9. PMID 24924557
- [Background] Tolsma V, Schwebel C, Azoulay E, Darmon M, Souweine B, Vesin A, Goldgran-Toledano D, Lugosi M, Jamali S, Cheval C, Adrie C, Kallel H, Descorps-Declere A, Garrouste-Orgeas M, Bouadma L, Timsit JF. Sepsis severe or septic shock: outcome according to immune status and immunodeficiency profile. Chest. 2014 Nov;146(5):1205-1213. doi: 10.1378/chest.13-2618. PMID 25033349
- [Background] Gunther SC, Schwebel C, Hamidfar-Roy R, Bonadona A, Lugosi M, Ara-Somohano C, Minet C, Potton L, Cartier JC, Vesin A, Chautemps M, Styfalova L, Ruckly S, Timsit JF. Complications of intravascular catheters in ICU: definitions, incidence and severity. A randomized controlled trial comparing usual transparent dressings versus new-generation dressings (the ADVANCED study). Intensive Care Med. 2016 Nov;42(11):1753-1765. doi: 10.1007/s00134-016-4582-2. Epub 2016 Oct 12. PMID 27734108